CLINICAL TRIAL: NCT02714608
Title: A PhaseⅡa, Placebo Parallel Control, Central Randomized, Double Blind, Dosage Exploring and Multi-Center Study to Evaluate the Efficacy and Safety of Ginsenoside H Dripping Pills in Patients With Advanced NSCLC (Syndrome Of Qi-Deficiency)
Brief Title: A Study of Ginsenoside H Dripping Pills for Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM0319
Record Dates: First submitted 2016-02-29; First posted 2016-03-21 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2016-03

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ginsenoside H dripping pills (Experimental): Drug: Ginsenoside H dripping pills. Dosage form:pill. Dosage :20pills ( only ginsenoside H dripping pills). Frequency:two times per day. Duration: until disease progression or death.
  Interventions: Drug: Ginsenoside H dripping pills
- Ginsenoside H dripping pills+Placebo (Experimental): Drug: Ginsenoside H dripping pills ,Placebo. Dosage form:pill. Dosage :20pills ( ginsenoside H dripping pills 10 pills and placebo 10 pills). Frequency:two times per day. Duration: until disease progression or death.
  Interventions: Drug: Ginsenoside H dripping pills+Placebo
- Placebo (Placebo Comparator): Drug: Placebo. Dosage form:pill. Dosage :20pills ( only placebo ). Frequency:two times per day. Duration: until disease progression or death.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginsenoside H dripping pills — Experimental: Ginsenoside H dripping pills. Dosage form:pill. Dosage :20pills ( only ginsenoside H dripping pills). Frequency:two times per day. Duration: until disease progression or death.
  Arms: Ginsenoside H dripping pills
Drug: Ginsenoside H dripping pills+Placebo — Experimental: Drug: Ginsenoside H dripping pills+Placebo. Dosage form:pill. Dosage :20pills ( ginsenoside H dripping pills 10 pills and placebo 10 pills). Frequency:two times per day. Duration: until disease progression or death.
  Arms: Ginsenoside H dripping pills+Placebo
Drug: Placebo — Placebo Comparator: Placebo. Dosage form:pill. Dosage :20pills ( only placebo ). Frequency:two times per day. Duration: until disease progression or death.
  Arms: Placebo

SUMMARY:
Ginsenoside H dripping pills is a kind of traditional Chinese medicine(TCM), This study is being conducted to evaluate the efficacy and safety of ginsenoside H dripping pills in patients with advanced (stage ⅢB/Ⅳ) Non-small Cell Lung Cancer (Syndrome Of Qi-Deficiency) and explore the optimal dosage

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically proven stage IIIB/IV NSCLC with a measurable lesions (including postoperative recurrence or metastasis)
2. The patients who can not be treated by surgical resection, conventional radiotherapy and chemotherapy or molecular targeted drugs treatment failure, not willing to accept, or intolerance to radiotherapy and chemotherapy or molecular targeted therapy.
3. The TCM Syndrome diagnosis of Qi-Deficiency.
4. Aged 18-75 years, both male and female.
5. ECOG performance status 0-2.
6. Expected to survive more than 3 months.
7. Joined in the test voluntarily and signed the Informed consent by GCP regulation.

Exclusion Criteria:

1. Liver and kidney damage(TBIL、ALT、AST is higher than the limit of normal value of 1.5 times, abnormal Cr).
2. Patients with significant cachexia.
3. Untreated symptomatic brain metastases.

4 .Allergic constitution, or for a variety of drug allergy.

5 .Combined with severe cardiovascular, hepatic, renal disease , pregnancy or breast-feeding women, psychopath.

6. Participated in other clinical trial within 3 months.

7. Treated by chemotherapy, radiotherapy or targeted therapy within 4 weeks.

8. Possible to be treated by chemotherapy, radiotherapy or targeted therapy during the study.

9. Not fit for the clinical trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | through study completion, an average of 1 year
  Evaluate progression free survival (PFS) in the 3 groups : 0 , every 8 weeks and the end of treatment

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 1 year
  Evaluate overall survival (OS) in the 3 groups
Time to progression(TTP) | through study completion, an average of 1 year
  Evaluate time to progression(TTP) in the 3 groups
Quality of Life | through study completion, an average of 1 year
  [0 , every 4 weeks and the end of treatment] To determine the quality of life by using the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scales.
Symptoms scores of TCM | through study completion, an average of 1 year
  0 , every 4 weeks and the end of treatment
Cancer-related fatigue | through study completion, an average of 1 year
  Evaluate the fatigue degree in the 3 groups using the Chinese version of Brief Fatigue Index (BFI-C): 0 , every 4 weeks and the end of treatment

OTHER OUTCOMES:
Blood routine test | through study completion, an average of 1 year
  0 , every 4 weeks during the period of 0 to 16 weeks, every 8 weeks after 16 weeks and the end of treatment
Urine routine test | through study completion, an average of 1 year
  0 , every 4 weeks during the period of 0 to 16 weeks, every 8 weeks after 16 weeks and the end of treatment
Hepatic function | through study completion, an average of 1 year
  0 , every 4 weeks during the period of 0 to 16 weeks, every 8 weeks after 16 weeks and the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, PhD, Study Director — Tasly Group, Co. Ltd.
Locations (9):
- China (9):
  - Guangdong Provincial Hospital of TCM, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong
  - Jiangsu Provincial Hospital of Integrated Chinese Traditional and Western Medicine, Nanjing, Jiangsu
  - Jing'an District Centre Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shuguang Hospital Affiliated with Shanghai University of TCM, Shanghai, Shanghai Municipality
  - West China Hospital ,Sichuan University, Chengdu, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No